CLINICAL TRIAL: NCT03110276
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Escalating Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of EYP001a in Healthy Male Subjects
Brief Title: Study Evaluating Safety, Tolerability and Pharmacokinetics of EYP001a in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYP001-C01; 2016-003035-37 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Planned single doses of 30 mg, 60 mg, 120 mg, 250 mg, 500 mg, and 800 mg, and planned multiple doses of 60 mg, 120 mg, 250 mg, and 500 mg, of EYP001a will be explored in this study. Subjects will be enrolled in dose escalation cohorts that will occur sequentially based upon review of safety and PK parameters.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EYP001a (Experimental)
  Interventions: Drug: EYP001a
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EYP001a — 10 mg and 100 mg capsules. Number of capsules to be ingested will depend on the dose cohort. Administered orally once daily. Single dose (SAD) or 14 days treatment (MAD).
  Other Names: EYP001
  Arms: EYP001a
Drug: Placebo — Placebo capsules, identical in appearance to the EYP001a 10 mg and 100 mg capsules.
  Arms: Placebo

SUMMARY:
The farnesoid X receptor (FXR) regulates hepatitis B virus replication through the bile acids pathway. EYP001a is a selective, synthetic FXR agonist under development for the treatment of hepatitis B.

This Phase 1 study is designed primarily to evaluate the single ascending dose (SAD) followed by a multiple ascending dose (MAD) safety, tolerability, and pharmacokinetics of EYP001a in healthy male subjects.

DETAILED DESCRIPTION:
This is a two-part, randomized, double-blind, placebo-controlled study. Healthy male subjects will be randomly assigned to receive EYP001a or placebo.

In the SAD part, up to 6 cohorts will receive EYP001a single doses of 30 mg, 60 mg, 120 mg, 250 mg, 500 mg, and 800 mg. In the MAD part, 4 cohorts will receive EYP001a doses of 60, 120, 250 and 500 mg, once daily for 14 days over 15-day period. Each cohort will include 6 active & 2 placebo subjects. Dose escalation will depend on evaluation of safety parameters.

Participation will include up to 21-day screening period followed by dosing period (1 to 15 days). A follow-up evaluation will occur at 6 ± 2 days post final dose.

Safety and tolerability will be assessed by monitoring adverse events, laboratory values, ECG parameters, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must satisfy all of the following inclusion criteria during screening to be enrolled in the study:

1. Subject has given voluntary written informed consent before performance of any study related procedure
2. Subject must be 18 to 50 years of age, inclusive at screening
3. Subject must have clinical chemistries, hematology, and urinalysis tests within normal, allowable limits (if out of range must be considered clinically significant to be exclusionary) and performed within 21 days of receiving first dose of study drug
4. Subject must have a body mass index of between 18 and 30 kg/m2 at screening
5. Subject must have weight > 60 kg at screening
6. Subject must have normal vital signs after 5 minutes resting in supine position at screening:

   * 95 mm Hg < systolic blood pressure < 140 mm Hg
   * 45 mm Hg < diastolic blood pressure < 90 mm Hg
   * 40 bpm < pulse rate < 90 bpm
7. Subject must have a normal 12-lead automatic ECG (incomplete right bundle branch block can be accepted): 120 ms < PR < 210 ms, QRS < 120 ms, corrected QT interval (QTc) (Fridericia) ≤ 450 msec at screening.
8. Agree to abstain from all medication, including non-prescription and prescription medication (including vitamins and natural or herbal remedies, e.g. St. John's Wort) for 21 days before the first study day until discharge from the study (end of post study medical).
9. Subject agrees to use condom from dosing through 90 days after the dose of study drug. Female partners of male subjects enrolled into this study are also recommended to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device,diaphragm, condom, or abstinence).

Exclusion Criteria:

-

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

1. A history of clinically significant gastrointestinal, especially peptic ulcerations, gastrointestinal bleeding, ulcerative colitis, cholecystectomy, Crohn's disease or Irritable Bowel Syndrome, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, especially those with a past history of depression, suicidal ideation or suicidal attempts, or cardiovascular disease or any other condition which, in the opinion of the principle investigator, would jeopardize the safety of the subject or impact the validity of the study results
2. Acute diarrhea or constipation in the 7 days before the predicted first study day. If screen occurs >7 days before first study day, this criterion will be determined on first study day. Diarrhea will be defined as the passage of liquid feces and/or a stool frequency of > 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
3. Donation or loss of more than 100 mL of blood within 60 days prior to the first drug administration
4. Regular alcohol consumption >21 units per week (1 Unit = 1⁄2 pint beer, 25 mL shot of 40% spirit or a 125 mL glass of wine)
5. Subject has a borderline or long QTc Fridericia interval as defined by screening readings of > 450
6. Subject has participated in a drug study within 60 days prior to the first drug administration in the current study
7. Subject has used any over-the-counter (OTC) medication, including vitamins, within 21 days prior to the study
8. Subject has used any prescription medication within 21 days prior to the study
9. Subject has been treated with any known P450 3A4 or 2D6 enzyme altering drugs within 30 days prior to the study
10. Subject smoking more than 5 cigarettes per day
11. Subject has sought advice from or been referred to a general practioner or counselor for abuse or misuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse, e.g. solvents
12. Subject has a positive blood screen for HIV, Hepatitis B surface antigen (HBsAg), and Hepatitis C Antibody and/or a positive urine screen for alcohol or drugs of abuse
13. Any current or previous use of drugs such as opiates, cocaine, ecstasy, or intravenous amphetamines

    - Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs-of-abuse test and have been abstinent from cannabis use for at least 3 months
14. Subject has an uncontrolled inter-current illness (i.e., active infection)
15. Subject has had major surgery within four weeks of study entry, or 12 months prior to study for gastrointestinal surgery.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is open to male subjects
Enrollment: 80 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects reported with adverse events, serious adverse events | 7 days (SAD) or 21 days (MAD)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of EYP001 | Days 1 & 2 (SAD and MAD). Days 14 & 15 (MAD)
  ng/mL
Time to reach maximum concentration after drug administration (Tmax) of EYP001 | Days 1 & 2 (SAD and MAD). Days 14 & 15 (MAD)
  hours
Area under the plasma concentration-time profile (AUCtau) of EYP001 | Days 1 & 2 (SAD and MAD). Days 14 & 15 (MAD)
  ng.h/mL
C4 (7α-hydroxy-4-cholesten-3-one) | Days 1 & 2 (SAD). Days 1, 7 & 15 (MAD)
  ng/mL
fibroblast growth factor 19 Fibroblast growth factor 19 (FGF19) | Days 1 & 2 (SAD). Days 1, 7 & 15 (MAD)
  pg/mL

IPD SHARING:
Plan to Share IPD: No